CLINICAL TRIAL: NCT03094039
Title: Initiation of Resuscitative Care While on Placental Circulation for Infants With Congenital Diaphragmatic Hernia - a Randomized Pilot Trial
Brief Title: Initiation of Resuscitation While Attached to the Cord With Congenital Diaphragmatic Hernia
Acronym: INSPIRE-CDH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient available for 18 months
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00069729
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilatory support while attached to the cord (Experimental): Infants will receive active resuscitative care (intubation and ventilation) using a specific designed platform for 120 seconds during delayed cord clamping. Then the cord will be clamped forgoing resuscitation care.
  Interventions: Procedure: Ventilatory support while attached to the cord
- Immediate cord clamping (Active Comparator): Infants will receive immediate cord clamping, transferred to the resuscitation table, intubated and mechanical ventilated according to our current Congenital Diaphragm Hernia protocol.
  Interventions: Procedure: Immediate cord clamping

INTERVENTIONS:
Procedure: Ventilatory support while attached to the cord — Infants will receive active resuscitative care (intubation and ventilation) using a specific designed platform for 120 seconds during delayed cord clamping. Then the cord will be clamped forgoing resuscitation care.
  Arms: Ventilatory support while attached to the cord
Procedure: Immediate cord clamping — Infants will receive immediate cord clamping, transferred to the resuscitation table, intubated and mechanical ventilated according to our current Congenital Diaphragm Hernia protocol.
  Arms: Immediate cord clamping

SUMMARY:
This study aims to measure the cardio-respiratory physiological consequences of initiating resuscitation during placental transfusion (PT) with an intact umbilical cord in infants with congenital diaphragmatic hernia (CDH). PT, mainly via delayed cord clamping, has been shown to offer a higher circulating blood volume, less need for blood transfusion, less need for inotropes in infants.

Currently infants with CDH receive immediate cord clamping (ICC) to facilitate immediate resuscitation including immediate intubation and mechanical ventilation.

With the development of a resuscitation platform (iNSPiRE), resuscitative care can now be commenced from birth in infants with CDH to benefit from PT.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants with an antenatal diagnosed CDH.

Exclusion Criteria:

* Severe antepartum or postpartum hemorrhage.
* Any obstetrical concern.
* Lack of parental consent.

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants with hypotension requiring inotropes | first 24 hours after birth
  Proportion of infants with hypotension requiring inotropes in the first 24 hours after birth in the neonatal intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No